CLINICAL TRIAL: NCT06910943
Title: A Phase 2b/3 Randomized Open-Label Dose-Selection Study With Open-Label Extension and Randomized Double-Blind, Placebo-Controlled Study With Open-Label Extension to Evaluate the Safety and Efficacy of Choline Chloride for Injection (Low Dose and High Dose) Versus Placebo in Adolescents and Adults With Intestinal Failure Receiving Long-Term Parenteral Support
Brief Title: Study of Choline Chloride for Injection in Adolescent and Adult Patients With Intestinal Failure Receiving Long Term Parenteral Support
Acronym: THRIVE-3
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Protara Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TARA-001-301
Record Dates: First submitted 2025-03-18; First posted 2025-04-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-10

CONDITIONS: Choline Deficiency; Liver Injury
Keywords: Intestinal Failure; Parenteral Nutrition; Parenteral Support; Choline Chloride; choline deficiency
MeSH Terms: conditions — Choline Deficiency; Intestinal Failure; Hyperphagia | interventions — Choline; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The Open-Label Dose Selection Phase will be open label, and the Double-Blind, Placebo-Controlled Phase will be double blind. The Open Label Extension Phase will be open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Open-Label, Dose-Selection: Dose 1 (Experimental)
  Interventions: Drug: Choline Chloride for Injection
- Open-Label, Dose-Selection: Dose 2 (Experimental)
  Interventions: Drug: Choline Chloride for Injection
- Open-Label, Dose-Selection: Dose 3 (Experimental)
  Interventions: Drug: Choline Chloride for Injection
- Double-Blind, Placebo-Controlled: High Dose (Experimental)
  Interventions: Drug: Choline Chloride for Injection
- Double-Blind, Placebo-Controlled: Low Dose (Experimental)
  Interventions: Drug: Choline Chloride for Injection
- Double-Blind, Placebo-Controlled: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Open Label Extension: High Dose (Experimental)
  Interventions: Drug: Choline Chloride for Injection
- Open Label Extension: Low Dose (Experimental)
  Interventions: Drug: Choline Chloride for Injection

INTERVENTIONS:
Drug: Choline Chloride for Injection — Intravenous use
  Arms: Double-Blind, Placebo-Controlled: High Dose; Double-Blind, Placebo-Controlled: Low Dose; Open Label Extension: High Dose; Open Label Extension: Low Dose; Open-Label, Dose-Selection: Dose 1; Open-Label, Dose-Selection: Dose 2; Open-Label, Dose-Selection: Dose 3
Drug: Placebo — Intravenous use
  Arms: Double-Blind, Placebo-Controlled: Placebo

SUMMARY:
TARA-001-301 is a Phase 2b/3 randomized Open-Label Dose-Selection study with an Open-Label Extension and randomized Double-Blind, Placebo-Controlled Study with Open-Label Extension to investigate the safety and efficacy of Choline Chloride for Injection (Low Dose and High Dose) versus Placebo in adolescents (ages 12 to < 18 years of age) and adults (≥ 18 years of age) with intestinal failure receiving long-term PS when oral or enteral nutrition is not possible, insufficient, or contraindicated.

Participants will be enrolled in one of 2 parts, each part will be followed by an open-label extension period of approximately a year.

Part 1: Open-Label Dose-Selection Phase Part 2: Double-Blind, Placebo-Controlled Phase

The purpose of the Open-Label Dose-Selection Phase is to evaluate the safety, tolerability, how Choline Chloride for Injection (study drug) is distributed in the body, and to select 2 of 3 doses for testing in the Double-Blind, Placebo-Controlled Phase.

The purpose of the Double-Blind, Placebo-Controlled Phase is to assess the safety of the study drug and how well the study drug works at the 2 selected dose levels.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female 12 years of age or older at the time of signing the informed consent
* Individuals who have voluntarily given written informed consent after the nature of the study has been explained according to applicable requirements, prior to study entry
* Individuals with intestinal failure receiving long-term PS when oral or enteral nutrition is not possible, insufficient, or contraindicated who are receiving stable PS at time of screening and for the duration of the study; Note: Long-Term PS = Participant must have been receiving PS for at least 6 months prior to screening and requiring PS at least 3 times per week
* Females of childbearing potential must have a negative urine pregnancy test at screening

Key Exclusion Criteria:

* Patients taking steatogenic medications for ≥ 12 weeks in the past 12 months; those taking any medicine that could affect the measurement of hepatic steatosis within 12 weeks prior to study entry
* Evidence of systemic active infection at the time of dosing
* Participants intending to take non-study drug choline supplements or choline-containing multivitamins during the course of the study
* Participants unwilling to limit alcohol intake to no more than 20/g a day for 24 hours prior to their screening visit and for the duration of the study
* Active malignancy (excluding basal cell skin tumor, low or very low risk prostate cancer, cervical carcinoma in situ and local resected cervical cancer)
* Clinically significant renal disease
* Low B12 or low serum folic acid levels that are less than the normal range
* Fulminant liver failure, with active bleeding and/or encephalopathy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Open-Label Dose-Selection Phase: PK of plasma free choline (Cmax) during Week 1 and Week 8 Visits | Week 1 to Week 8
  Cmax = maximum concentration
Open-Label Dose-Selection Phase: Open-Label Dose-Selection Phase: PK of plasma free choline (Tmax) during Week 1 and Week 8 Visits | Week 1 to Week 8
  Tmax = time of maximum concentration
Open-Label Dose-Selection Phase: PK of plasma free choline (AUC(0-TAU)) during Week 1 and Week 8 Visits | Week 1 to Week 8
  AUC = area under the curve, AUC(0-TAU) = AUC at end of dosing
Open-Label Dose-Selection Phase: Change from Baseline in plasma free choline concentrations at Week 8 | Week 1 to Week 8
Open-Label Dose-Selection Phase and Double-Blind, Placebo-Controlled Phase, Open-Label Extension Phase: Incidence and severity of TEAEs Incidence of TESAEs | Week 1 to Week 64
  TEAE = treatment emergent adverse event, TESAE = treatment emergent serious adverse event
Double-Blind, Placebo-Controlled Phase: Change from Baseline in peak plasma free choline concentrations (Cmax) at Week 8 in participants receiving Choline Chloride for Injection versus Placebo | Week 1 to Week 8
  Tmax = time of maximum concentration
Open-Label Extension Phase: Participants from Open-Label Dose-Selection Phase: Percentage of participants with plasma free choline concentrations of ≥ 9.5 nmol/mL at Week 64 | Week 64
Open-Label Extension Phase: Percentage of participants maintaining plasma free choline concentrations of ≥ 9.5 nmol/mL at Week 8 and Week 64 (ie, both timepoints) | Week 8 to Week 64
Open-Label Extension Phase: Participants from Double-Blind, Placebo-Controlled Phase: % with plasma free choline concentrations of ≥9.5 nmol/mL at Week 64 | Week 1 to Week 64
Open-Label Extension Phase: Participants from Double-Blind Placebo-Controlled Phase: % maintaining plasma free choline concentrations of ≥ 9.5 nmol/mL at Week 8, Week 24 and Week 64 for participants who previously received Choline Chloride for Injection | Week 8 to Week 64

SECONDARY OUTCOMES:
Open-Label Dose-Selection Phase: Change from Baseline to Week 8 in ALP, AST, ALT, GGT, VLDL, total bilirubin, direct bilirubin levels, CPK, homocysteine and albumin levels | Week 1 to Week 8
  ALP = alkaline phosphatase, AST = aspartate aminotransferase, ALT = alanine transaminase, GGT = gamma-glutamyl transpeptidase, VLDL = very low-density lipoprotein, CPK = creatine phosphokinase
Open-Label Dose-Selection Phase: Triplicate QTc measurements collected during Week 1 and Week 8, and changes from pre-infusion QTc at Week 1 to all post-baseline timepoints | Week 1 to Week 8
  QTc = QT corrected for heart rate
Open-Label Dose-Selection Phase: Percentage of participants achieving plasma free choline concentration Cmax ≥ 9.5 nmol/mL at Week 8 | Week 1 to Week 8
  Cmax = maximum concentration
Open-Label Dose-Selection Phase: Percentage of participants maintaining plasma free choline concentration Cmax ≥ 9.5 nmol/mL at Week 8 | Week 1 to Week 8
  Cmax = maximum concentration
Open-Label Dose-Selection Phase: Change from Baseline to Week 8 in height, weight and BMI | Week 1 to Week 8
  BMI = body mass index Weight and height will be combined to report BMI in kg/m^2
Open-Label Dose-Selection Phase: Percentage of participants with no worsening of steatosis from Baseline to Week 8 as measured by MRI-PDFF | Week 1 to Week 8
  MRI-PDFF = magnetic resonance imaging-estimated proton density fat fraction
Open-Label Dose-Selection Phase: Percentage of participants with any improvement of steatosis from Baseline to Week 8 as measured by MRI-PDFF | Week 1 to Week 8
  MRI-PDFF = magnetic resonance imaging-estimated proton density fat fraction
Double-Blind, Placebo-Controlled Phase: Change from Baseline and Week 8 in peak plasma free choline concentrations (Cmax) at Week 24 in participants receiving Choline Chloride for Injection versus Placebo | Week 1 to Week 24
  Tmax = time of maximum concentration
Double-Blind, Placebo-Controlled Phase: Percentage of participants achieving plasma free choline concentration Cmax ≥ 9.5 nmol/mL at Week 8 | Week 1 to Week 8
  Cmax = maximum concentration
Double-Blind, Placebo-Controlled Phase: Percentage of participants maintaining plasma free choline concentration Cmax ≥ 9.5 nmol/mL at Week 8 and Week 24 (ie, through Week 24) | Week 1 to Week 24
  Cmax = maximum concentration
Double-Blind, Placebo-Controlled Phase: Change from Baseline to Week 8 and Week 24 in height, weight and BMI | Week 1 to Week 24
  BMI = body mass index Weight and height will be combined to report BMI in kg/m^2
Double-Blind, Placebo-Controlled Phase: Change from Baseline to Week 8 and Week 24 in ALP, AST, ALT, GGT, VLDL, total bilirubin, direct bilirubin levels, CPK, homocysteine and albumin levels | Week 1 to Week 24
  ALP = alkaline phosphatase, AST = aspartate aminotransferase, ALT = alanine transaminase, GGT = gamma-glutamyl transpeptidase, VLDL = very low-density lipoprotein, CPK = creatine phosphokinase
Double-Blind, Placebo-Controlled Phase: Percentage of participants with no worsening of steatosis from Baseline to Week 24 as measured by MRI-PDFF | Week 1 to Week 24
  MRI-PDFF = magnetic resonance imaging-estimated proton density fat fraction
Double-Blind, Placebo-Controlled Phase: Percentage of participants with any improvement of steatosis from Baseline on MRI-PDFF at Week 24 | Week 1 to Week 24
  MRI-PDFF = magnetic resonance imaging-estimated proton density fat fraction
Double-Blind, Placebo-Controlled Phase: Percentage of participants with no worsening in fibrosis grade from Baseline to Week 24, as measured by MRE and ELF test | Week 1 to Week 24
  MRE = magnetic resonance elastography, ELF = enhanced liver fibrosis
Double-Blind, Placebo-Controlled Phase: Percentage of participants with improvement in fibrosis grade from Baseline to Week 24, as measured by MRE and ELF test | Week 1 to Week 24
  MRE = magnetic resonance elastography, ELF = enhanced liver fibrosis
Double-Blind, Placebo-Controlled Phase: Percentage of participants with improvement of steatosis from Baseline on MRI-PDFF with improvement of ALP from Baseline to Week 24 | Week 1 to Week 24
  MRI-PDFF = magnetic resonance imaging-estimated proton density fat fraction, ALP = alkaline phosphatase
Double-Blind, Placebo-Controlled Phase: Percentage of participants with improvement of steatosis from Baseline on MRI-PDFF with improvement of ALT or AST from Baseline to Week 24 | Week 1 to Week 24
  MRI-PDFF = magnetic resonance imaging-estimated proton density fat fraction, ALT = alanine transaminase, AST = aspartate aminotransferase
Double-Blind, Placebo-Controlled Phase: Assessment of Quality of Life based on CLDQ at Baseline and Week 24 | Week 1 to Week 24
  CLDQ = chronic liver disease questionnaire
Double-Blind, Placebo-Controlled Phase: Assessment of Quality of Life based on PGIS at Baseline and PGIC at Week 24 | Week 1 to Week 24
  PGIC = patient global impression of change
Open-Label Extension Phase: Participants from Open-Label Dose-Selection Phase: Change from Baseline (Week 1) to Week 64 in ALP, AST, ALT, GGT, VLDL, total bilirubin, direct bilirubin levels, CPK, homocysteine and albumin levels | Week 1 to Week 64
  ALP = alkaline phosphatase, AST = aspartate aminotransferase, ALT = alanine transaminase, GGT = gamma-glutamyl transpeptidase, VLDL = very low-density lipoprotein, CPK = creatine phosphokinase
Open-Label Extension Phase: Double-Blind, Placebo-Controlled Phase: Change from W1 to W64 in Choline Chloride for Injection group, and change from W24 to W64 in Placebo group in ALP, AST, ALT, GGT, VLDL, TBIL, DBil levels, CPK, homocysteine and albumin | Week 1 to Week 64
  ALP = alkaline phosphatase, AST = aspartate aminotransferase, ALT = alanine transaminase, GGT = gamma-glutamyl transpeptidase, VLDL = very low-density lipoprotein, CPK = creatine phosphokinase, TBIL = total bilirubin, DBil = direct bilirubin
Open-Label Extension Phase: Participants from Open-Label Dose-Selection Phase Change from Baseline (Week 1) to Week 64 in height, weight and BMI | Week 1 to Week 64
  BMI = body mass index Weight and height will be combined to report BMI in kg/m^2
Open-Label Extension Phase: Participants from Double-Blind, Placebo-Controlled Phase: Change from W1 to W64 for participants in Choline Chloride for Injection group, and change from W24 to W64 for participants in Placebo group in height, weight and BMI | Week 1 to Week 64
  BMI = body mass index Weight and height will be combined to report BMI in kg/m^2
Open-Label Extension Phase: Participants from Open-Label Dose-Selection Phase: Percentage of participants with no worsening of steatosis as measured by MRI-PDFF from Baseline (Week 1) to Week 64 | Week 1 to Week 64
  MRI-PDFF = magnetic resonance imaging-estimated proton density fat fraction
Open-Label Extension Phase: Participants from Open-Label Dose-Selection Phase: Percentage of participants with improvement of steatosis as measured by MRI-PDFF from Baseline (Week 1) to Week 64 | Week 1 to Week 64
  MRI-PDFF = magnetic resonance imaging-estimated proton density fat fraction
Open-Label Extension Phase: Participants from Double-Blind, Placebo-Controlled Phase: % of participants with no worsening of steatosis measured by MRI-PDFF from W1 to W64 in Choline Chloride for Injection group, and from W24 to W64 in Placebo group | Week 1 to Week 64
  MRI-PDFF = magnetic resonance imaging-estimated proton density fat fraction
Open-Label Extension Phase: Participants from Double-Blind, Placebo-Controlled Phase: % of participants with improvement of steatosis measured by MRI-PDFF from W1 to W64 in Choline Chloride for Injection group, and from W24 to W64 in Placebo group | Week 1 to Week 64
  MRI-PDFF = magnetic resonance imaging-estimated proton density fat fraction
Open-Label Extension Phase: Double-Blind, Placebo-Controlled Phase: % of participants with no worsening in fibrosis grade measured by MRE and ELF test from W1 to W64 in Choline Chloride for Injection group, and from W24 to W64 in Placebo group | Week 1 to Week 64
  MRE = magnetic resonance elastography, ELF = enhanced liver fibrosis
Open-Label Extension Phase: Participants from Double-Blind, Placebo-Controlled Phase: % of participants with improvement in fibrosis measured by MRE and ELF test from W1 to W64 in Choline Chloride for Injection group, and W24 to W64 in Placebo group | Week 1 to Week 64
  MRE = magnetic resonance elastography, ELF = enhanced liver fibrosis
Open-Label Extension Phase: Participants from Double-Blind Placebo-Controlled Phase: Assessment of QOL based on CLDQ at Week 64 | Week 64
  QOL = quality of life, CLDQ = chronic liver disease questionnaire
Open-Label Extension Phase: Participants from Double-Blind Placebo-Controlled Phase: Assessment of QOL based on PGIC at Week 64 | Week 64
  QOL = quality of life, PGIC = patient global impression of change

CONTACTS AND LOCATIONS:
Overall Officials: Chief Scientific Operations Officer, Study Director — Protara Therapeutics
Locations (14):
- United States (4):
  - University of Colorado School of Medicine, Aurora, Colorado
  - Columbia University Medical Center/ New York Presbyterian Hospital, New York, New York
  - Duke Clinic - Abdominal Transplant Research Office, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
- University Hospitals Leuven, Campus Gasthuisberg, Leuven, Belgium
- Denmark (2):
  - Aalborg University Hospital, Department of Medical Gastroenterology, Aalborg
  - Rigshospitalet - University Hospital Copenhagen, Copenhagen
- France (3):
  - Beaujon Hospital - APHP, Clichy
  - Rennes University Hospital Center - Pontchaillou Site, Rennes
  - CHRU Nancy - Barbois Hospital, Vandœuvre-lès-Nancy
- Germany (2):
  - Charite - University Hospital Berlin, Berlin
  - University Duisburg-Essen, University Hospital Essen, Essen
- Poland (2):
  - M. Pirogow Provincial Specialized Hospital in Lodz, Nutritional Treatment Center, Lodz
  - Czerniakowski Hospital Sp. z o.o. (LCC), Warsaw

IPD SHARING:
Plan to Share IPD: No